CLINICAL TRIAL: NCT05063396
Title: The Efficacy and Safety of Opioid-free Anesthesia(OFA) for Non-small-cell Lung Cancer Resection and Its Underlying Clinical Value: a Prospective Study
Brief Title: OFA in Thoracic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OFAbywang
Record Dates: First submitted 2021-05-10; First posted 2021-10-01 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Thoracic Cancer
Keywords: opioid free anesthesia; non small cell lung caner

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- opioid free anesthesia (Active Comparator): opioid free anesthesia
  Interventions: Procedure: opioid free anesthesia
- Opioid-sparing anesthesia (Placebo Comparator): Opioid-sparing anesthesia
  Interventions: Procedure: Opioid-sparing anesthesia

INTERVENTIONS:
Procedure: opioid free anesthesia — Instead of use of large amount of opioids for intraoperative stress response and postoperative pain controlling, during the whole perioperative period patients received no opioid at all. intravenous local anesthetics and thoracic epidural were used.
  Arms: opioid free anesthesia
Procedure: Opioid-sparing anesthesia — patients will receive opioid-sparing anesthesia protocol with minimal intraoperative sufentanil, remifentanil and epidural hydromorphone.
  Arms: Opioid-sparing anesthesia

SUMMARY:
to investigate the efficacy and safety of opioid-free anesthesia for non-small-cell lung cancer resection and its underlying clinical value

DETAILED DESCRIPTION:
Opioids used to have its irreplaceable role in standard opioid-based anesthesia, yet with the help of hypnotics, local anesthetics, anti-inflammatory drugs, α-2 agonists and epidural techniques, opioid-free anesthesia (OFA) has been proved to be safe and feasible for non-cardiac major surgeries. Opioid-sparing anesthesia (OSA) is encouraged by the needs of enhanced recovery and recommended by the latest guidelines for anesthesia of lung surgery. According to previous studies, both opioid-sparing and opioid-free anesthesia would reduce the incidence of opioid-related adverse events and speed up the postoperative recovery to some extent, yet no studies ever are dedicated to compare these two different techniques.

ELIGIBILITY:
Inclusion Criteria:

* going through thoracoscopic lung surgery including lobectomy, segmentectomy, single or multiple wedge resection, and two of the above procedures combined;
* able to complete the pain scoring face-to-face;
* no cognitive dysfunction or history of anesthetic drug allergy;
* ASA grade I-II

Exclusion Criteria:

-psychological disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
acute postoperative pain scores | day1 postoperation
  visual analog scale was used
acute postoperative pain scores | day2 postoperation
  visual analog scale was used
occurrence of postoperative opioid-related adverse events | day1 postoperation
  occurrence of postoperative opioid-related adverse events
occurrence of postoperative opioid-related adverse events | day2 postoperation
  occurrence of postoperative opioid-related adverse events

SECONDARY OUTCOMES:
relapse free survival and overall survival | within 5 years
  relapse free survival and overall survival
occurrence of episodes of postoperative pain (VAS ≥4) | within 48hours
  occurrence of episodes of postoperative pain (VAS ≥4)
PCEA bolus consumption | within 48hours
  PCEA bolus consumption
need for rescue intravenous opioids or any type of painkiller | within 48hours
  need for rescue intravenous opioids or any type of painkiller
hospital length of stay and total hospital expenses | within 10days
  hospital length of stay and total hospital expenses
Pathologic results and TNM rating | within one month
  Pathologic results and TNM rating

CONTACTS AND LOCATIONS:
Overall Officials: Changhong Miao, Study Chair — Shanghai Zhongshan Hospital
Locations (2):
- China (2):
  - 180 Fenglin Road, Shanghai
  - Zhongshan Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devine G, Cheng M, Martinez G, Patvardhan C, Aresu G, Peryt A, Coonar AS, Roscoe A. Opioid-Free Anesthesia for Lung Cancer Resection: A Case-Control Study. J Cardiothorac Vasc Anesth. 2020 Nov;34(11):3036-3040. doi: 10.1053/j.jvca.2020.05.022. Epub 2020 May 27. PMID 32682739
- [Background] Bello M, Oger S, Bedon-Carte S, Vielstadte C, Leo F, Zaouter C, Ouattara A. Effect of opioid-free anaesthesia on postoperative epidural ropivacaine requirement after thoracic surgery: A retrospective unmatched case-control study. Anaesth Crit Care Pain Med. 2019 Oct;38(5):499-505. doi: 10.1016/j.accpm.2019.01.013. Epub 2019 Feb 5. PMID 30731138
- [Derived] Wang S, Li Y, Liang C, Han X, Wang J, Miao C. Opioid-free anesthesia reduces the severity of acute postoperative motion-induced pain and patient-controlled epidural analgesia-related adverse events in lung surgery: randomized clinical trial. Front Med (Lausanne). 2023 Nov 6;10:1243311. doi: 10.3389/fmed.2023.1243311. eCollection 2023. PMID 38020116